CLINICAL TRIAL: NCT04514120
Title: Development and Validation of a Descriptive and Clinically Relevant Postoperative Endoscopic Sinus Scoring System
Brief Title: Alsaleh-Javer Endoscopic Sinus Score (AJESS) System
Acronym: AJESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Assistant Clinical Professor, St. Paul's Hospital, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H20-02108
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Chronic Rhinosinusitis; Endoscopic score
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: This mixed-methods clinical study of patients with CRS includes both a cross-sectional arm (single participant encounter with stable patients, n=100) and a second prospective aspect (3 participant encounters with patients experiencing CRS exacerbation, n=30)
Masking Description: This is not a blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stable CRS (Experimental): Patients diagnosed with Chronic Rhinosinusitis including those with or without nasal polyposis and/or with Allergic Fungal Rhinosinusitis and stable condition
  Interventions: Other: AJESS scoring process
- Non-stable CRS (Experimental): Patients diagnosed with Chronic Rhinosinusitis including those with or without nasal polyposis and with Allergic Fungal Rhinosinusitis who are experiencing an exacerbation
  Interventions: Other: AJESS scoring process

INTERVENTIONS:
Other: AJESS scoring process — We will collecto endoscopic pictures from stable and non stable participants. Pictures will be taken for each sinus, olfactory cleft, and middle meatus in private clinical exam rooms. For each anatomic site [left middle meatus (LMM), left ethmoid sinus (LES), left frontal sinus (LFS), left maxillary sinus (LMS), left olfactory cleft (LOC), left sphenoid sinus (LSS), right middle meatus (RMM), right ethmoid sinus (RES), right frontal sinus (RFS), right maxillary sinus (RMS), right olfactory cleft (ROC), right sphenoid sinus (RSS)], numerical scores describe edema or polyposis while alphabetical scores, in lower case or upper case corresponding to severity, describe CRS features: crusting, synechiae, purulence, mucus, recirculation, and ostial narrowness.

SUMMARY:
Several endoscopic scores have been developed to assess Chronic Rhinosinusitis severity like the Modified Lund-Kennedy (MLK). This is a simple score only based on endoscopic signs. We proposed a more descriptive Alsaleh-Javer Endoscopic Sinus Score (AJESS) system which assesses all sinuses and nasal passages based on participant's severity of symptoms too. This would be a more reliable and clinically valid CRS endoscopic score. We aim to study thE AJESS system in 100 participants with stable CRS and 30 participants CRS who are experiencing an exacerbation (worsening of CRS).

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a prevalent inflammatory disorder of the nasal passages and sinuses associated with detrimental effects on quality of life and productivity as well as billions of dollars in healthcare expenses and lost productivity each year. Numerous endoscopic scoring systems have been developed to assess CRS disease severity such as the popular Modified Lund-Kennedy (MLK) score which assesses sinus cavities only based on 3 criteria (polyps, edema, and discharge) with small 0-2 integer scales. Yet, such systems at best have reported good to moderate reliabilities and weak to no correlation with patient-reported outcome measures (PROMs) which should motivate further research to develop a more reliable and clinically valid CRS endoscopic scoring system, especially one which can better align the observed endoscopic signs of disease with the severity of symptoms reported by patients. In this study we propose a more descriptive Alsaleh-Javer Endoscopic Sinus Score (AJESS) system which assesses all sinuses and nasal passages with a numerical score of inflammation severity, alphabetical score for presence of CRS features, and an aggregated numerical score of overall disease severity. Our mixed-methods clinical study of 100 stable post-operative CRS patients and 30 post-operative CRS patients experiencing an exacerbation who are visiting St. Paul's Sinus Centre will gather both cross-sectional (1 visit, CRS stable) and prospective (2 follow-up visits approximately 2-4 weeks apart each, CRS flares) clinical data including two PROMs (SNOT-22, VAS) and an objective olfactory sensation test (Sniffin' Sticks TDI Score) to assess AJESS and MLK scores in terms of inter-rater reliability, test-retest reliability, correlation with clinical data, and responsiveness to changes in clinical data. Pending validation and head-to-head analysis with the MLK score, the AJESS system may be a more reliable and valid endoscopic scoring system for clinical practice and outcomes research in CRS.

Study goals and objectives

1. Assess the test-retest and inter-rater reliability of the AJESS and MLK scores.
2. Assess the correlation of AJESS and MLK scores with cross-sectional PROMs (SNOT-22, VAS) and Sniffin' Sticks TDI Score
3. Assess the reactivity of AJESS and MLK scores with prospective PROMs (SNOT-22, VAS) in patients experiencing CRS exacerbations

Research design

Participants visiting St. Paul's Sinus Centre who meet inclusion criteria and no exclusion criteria who are stable (N=100) and who are experiencing an exacerbation (N=30) will be approached at random and consented to the study. Encounters are expected to be 30 minutes each and participants experiencing a CRS or AFRS exacerbation will be expected to present for follow-up after 3 weeks (+/- 1 week) intervals for a second and a third encounter until their exacerbation are settled. The first encounter will collect relevant clinical data, endoscopic photos of 10 anatomic sites, patient-reported outcomes measures (PROMs, eg.SNOT-22, VAS) and olfactory sense test results (Sniffin' Sticks TDI score). Subsequent visits for exacerbated participants will collect the same endoscopic photos, PROMs and olfactory sense test results.

ELIGIBILITY:
Inclusion Criteria:

* Are over 19 years old
* Patients diagnosed with Chronic Rhinosinusitis including those with or without nasal polyposis and with Allergic Fungal Rhinosinusitis
* Post-operative patients

Exclusion Criteria:

* Have a sinonasal neoplasm
* Have syndromic sinusitis e.g. cystic fibrosis or vasculitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Test-retest and inter-rater reliability of the AJESS compare to MLK scores. | Baseline

SECONDARY OUTCOMES:
Change in the SNOT-22 between the AJESS and MLK in stable participants | Baseline
  The Sinonasal Outcome Test includes 22 questions about symptoms and social/emotional consequences of participant's nasal disorder. Participants will be asked to rate their problems as they have been over the past two weeks. A score will be given out of 110 where a higher score indicates a worse outcome.
Change in the VAS between the AJESS and MLK score in stable participants | Baseline
  Pain and discomfort (Visual Analog Scale): The visual analog score describes subjective pain and discomfort levels experienced by the participant about the sinus disease overall The scoring would be from 0 or No At All Severe/Doesn't Bother me at All to 10 Extremely Severe/ Bothers me very much
Change in the Sniffin' Stick TDI between the AJESS and MLK score in stable participants | Baseline
  Sniffn' Sticks is a type of test to assess your sense of smell by using various scented pens. The threshold and identification tests will be performed. A score will be given out of 32 with a lower score indicating a worse outcome/sense of smell.

OTHER OUTCOMES:
Change in SNOT-22 between the AJESS and MLK score in exacerbated patients | Baseline and 3 weeks
  The Sinonasal Outcome Test includes 22 questions about symptoms and social/emotional consequences of participant's nasal disorder. Participants will be asked to rate their problems as they have been over the past two weeks. A score will be given out of 110 where a higher score indicates a worse outcome.
Change in SNOT-22 between the AJESS and MLK score in exacerbated patients | Baseline and 6 weeks
  The Sinonasal Outcome Test includes 22 questions about symptoms and social/emotional consequences of participant's nasal disorder. Participants will be asked to rate their problems as they have been over the past two weeks. A score will be given out of 110 where a higher score indicates a worse outcome.
Change in the VAS between the AJESS and MLK score in exacerbated participants | Baseline and 3 weeks
  Pain and discomfort (Visual Analog Scale): The visual analog score describes subjective pain and discomfort levels experienced by the participant about the sinus disease overall The scoring would be from 0 or No At All Severe/Doesn't Bother me at All to 10 Extremely Severe/ Bothers me very much
Change in the VAS between the AJESS and MLK score in exacerbated participants | Baseline and 6 weeks
  Pain and discomfort (Visual Analog Scale): The visual analog score describes subjective pain and discomfort levels experienced by the participant about the sinus disease overall The scoring would be from 0 or No At All Severe/Doesn't Bother me at All to 10 Extremely Severe/ Bothers me very much